CLINICAL TRIAL: NCT03301844
Title: Randomized, Controlled Study With a Closed Sequential Design to Compare the Efficacy, Safety and Patient Satisfaction of Blephapad Combo vs. Standard Treatment for Eyelid Cleansing in Patients Affected by Bilateral Posterior Blepharitis.
Brief Title: To Compare Blephapad Combo vs Standard Treatment for Eyelid Cleansing in Bilateral Posterior Blepharitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLEPHA 01-2017
Record Dates: First submitted 2017-08-02; First posted 2017-10-04 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-11

CONDITIONS: Bilateral Blepharitis (Disorder)

STUDY DESIGN:
Intervention Model Description: A randomized, controlled study with a closed sequential design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study treatment (Experimental): Blephapad Combo twice daily for one month. Blephapad is a disposable wet wipe containing Hy-Ter® solution (sodium hyaluronate acid and 4-terpineol), aloe, natural anti-inflammatories and antiseptics.
  Interventions: Combination Product: Blephapad Combo
- Standard treatment (Other): Wet, warm gauze twice daily for one month.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Combination Product: Blephapad Combo — Blephapad Combo is used to cleanse, soften, sooth and decongest inflamed eyelids and cilia.
  The combo also presents an applicator with a heatable tablet that is applied to the eyelid in order to clean and open occluded Meibomian glands, thereby allowing the production of lipids necessary for a healthy tear film. The heatable tablet is to be used prior to cleansing with Blephapad wipes.
  Arms: Study treatment
Other: Standard treatment — Standard treatment, twice daily for one month, consisting in eyelid hygiene using wet, warm gauze.
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy of, and patient satisfaction with Blephapad Combo in the treatment of posterior blepharitis.

DETAILED DESCRIPTION:
Blepharitis is the most common condition in patients seeking an eye examination due to discomfort or eye irritation. Treatment of blepharitis is recommended even in mild cases as chronic inflammation may cause permanent damage to the Meibomian glands.

Each eye of each patient represents an experimental unit. Each patient will apply Blephapad Combo to one eye and standard treatment to the other eye in accordance with the randomization procedure.

The aim of this randomized, controlled study with a closed sequential design is to evaluate versus standard treatment the efficacy of, and patient satisfaction with Blephapad Combo in the treatment of posterior blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* Male or female
* Diagnosis of bilateral posterior blepharitis
* Written informed consent of patient

Exclusion Criteria:

* Treatment with topical ophthalmic drugs (artificial tears allowed)
* Ocular surgery in the previous 6 months
* Pregnant or breastfeeding women
* Alcohol abuse
* Psychiatric disorders
* Cognitive impairment that could affect evaluation of preferences
* Participation in other clinical studies in the last month
* Hypersensitivity to one or more components of the study products

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Scorcia, Principal Investigator — A.O.U. Policlinico Mater Domini
Locations (1):
- A.O.U. Policlinico Mater Domini, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Luca V, Carnevali A, Carnovale Scalzo G, Piccoli G, Bruzzichessi D, Scorcia V. Efficacy and Safety of Wet Wipes Containing Hy-Ter(R) Solution Compared with Standard Care for Bilateral Posterior Blepharitis: A Preliminary Randomized Controlled Study. Ophthalmol Ther. 2019 Jun;8(2):313-321. doi: 10.1007/s40123-019-0182-x. Epub 2019 Mar 30. PMID 30929188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2017 and January 2018 at the Ophthalmology Unit of the Magna Graecia University of Catanzaro in Italy
Pre-assignment Details: During a 2-week run-in period starting at Visit 1, and after the patient has provided informed consent, the Investigator will collect demographic data and medical history and perform a physical examination of the patient.
Units Other Than Participants: eyes
Groups:
- Study Treatment: Blephapad Combo twice daily for one month. Blephapad is a disposable wet wipe containing Hy-Ter® solution (sodium hyaluronate acid and 4-terpineol), aloe, natural anti-inflammatories and antiseptics.
  Blephapad Combo: Blephapad Combo is used to cleanse, soften, sooth and decongest inflamed eyelids and cilia.
  The combo also presents an applicator with a heatable tablet that is applied to the eyelid in order to clean and open occluded Meibomian glands, thereby allowing the production of lipids necessary for a healthy tear film. The heatable tablet is to be used prior to cleansing with Blephapad wipes.
Period: Overall Study
Arm/Group | Study Treatment | Standard Treatment
Started | 19; 19 eyes (Each patient apply the Blephapad Combo wipes to one eye and standard treatment to the other eye.) | 19; 19 eyes (Each patient apply the Blephapad Combo wipes to one eye and standard treatment to the other eye.)
Completed | 18; 18 eyes | 18; 18 eyes
Not Completed | 1; 1 eyes | 1; 1 eyes
Not completed — suspected colon cancer | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients aged > 40 years with symmetrical bilateral posterior blepharitis. Each eye represented a single experimental unit.
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Treatment | Standard Treatment | Total
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (eyes) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: One patient was excluded due to suspected colon cancer.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 5 | 10
    >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient was excluded due to suspected colon cancer.
  years | 66.9 (9.03) | 66.9 (9.03) | 66.9 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient was excluded due to suspected colon cancer
  Participants
    Female | 9 | 9 | 18
    Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient was excluded due to suspected colon cancer.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 18 | 18 | 36
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: One patient was excluded due to suspected colon cancer.
  participants
    Italy | 18 | 18 | 18
Meibomian Gland Dysfunction (MGD) at baseline (visit 2) [Mean (Standard Deviation); unit: score on a scale] — The total score of the meibomian gland dysfunction (MGD) grading scale was automatically computed by the system as the sum of the six sub-scores (Lid margin findings of vascularity, Plugging of gland orifices, Lid margin irregularity, Lid margin thickening, Partial glands and Gland dropout), ranging from 0 to 15. The first four parameters were evaluated using photographic images of anterior segments, while the last two were evaluated using infrared images of the meibomian glands. Higher scores implied a worse meibomian gland condition while lower scores were correlated to a better condition. Population: One patient was excluded due to suspected colon cancer.
  score on a scale | 9.17 (2.64) | 9.39 (2.73) | 9.28 (2.65)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of the Total Score of the Grading Scales for Meibomian Gland Dysfunction (MGD)
Description: The total score of the meibomian gland dysfunction (MGD) grading scale was automatically computed by the system as the sum of the six sub-scores (i.e. Lid margin findings of vascularity, Plugging of gland orifices, Lid margin irregularity, Lid margin thickening, Partial glands and Gland dropout), ranging from 0 to 15, where higher values rapresent a worse outcome.
  The first four parameters were evaluated using photographic images of anterior segments, while the last two were evaluated using infrared images of the meibomian glands Based on the percentage change from baseline to week 4 of the total score of MGD score, Investigators will choose which of the two eyes had a better change of clinical features.
Time Frame: from baseline to week 4
Population: patients with symmetrical bilateral posterior blepharitis
Measure: Mean (Standard Deviation); unit: percentage of change in the total score
Arm/Group | Study Treatment | Standard Treatment
Number analyzed (Participants) | 18 | 18
percentage of change in the total score | -38.5 (21.3) | -29.9 (17.6)

2. Secondary Outcome: Change of the Total Score of the Grading Scales for Meibomian Gland Dysfunction (Improved vs Not Improved)
Description: For each eye change from baseline to week 4 in the total score of Meibomian Gland Dysfunction was also expressed as one of the following outcomes:
  1. Eye on Blephapad Combo: Improved-Eye on Standard: Improved
  2. Eye on Blephapad Combo: Improved-Eye on Standard: NOT Improved
  3. Eye on Blephapad Combo: NOT Improved-Eye on Standard: Improved
  4. Eye on Blephapad Combo: NOT Improved-Eye on Standard: NOT Improved
  The total score was automatically computed by the system as the sum of the six sub-scores (i.e. Lid margin findings of vascularity, Plugging of gland orifices, Lid margin irregularity, Lid margin thickening, Partial glands and Gland dropout), ranging from 0 to 15 (higher values rapresent a worse outcome).If the change of the total score was positive or equal to 0 the specific eye was referred as "NOT improved",on the contrary if the change of the total score resulted negative the specific eye was referred as "Improved". For each patient the results on the two eyes were combined.
Time Frame: From Visit 2 (baseline) to Visit 3 (week 4)
Population: Patiens with symmetrical bilateral posterior blepharitis who applied treatment at least once in one eye and had a baseline evaluation of the primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment | Standard Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Eye improved | 16 | 15
  Eye NOT improved | 1 | 2
  Missing | 1 | 1

3. Secondary Outcome: Number of Patients Preferring the Standard or the Study Treatment (i.e. Answers to a Specific Question on Patient Preference: Study Drug vs. Standard Treatment)
Description: At the end of study patients was asked to state their preference on the treatments used.
Time Frame: at Visit 3 (week 4)
Population: Patiens with symmetrical bilateral posterior blepharitis who applied treatment at least once in one eye and had a baseline evaluation of the primary efficacy endpoint. One patient didn't express the preference therefore 17 patients were considered.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment | Standard Treatment
Number analyzed (Participants) | 17 | 17
Participants | 12 | 5
Statistical Analysis 1: Comparison: Study Treatment vs Standard Treatment; Test type: Superiority; p = 0.071, Chi-squared; Patient preference for one of the two treatments at Visit 3 was presented overall in terms of number and percentage of patients preferring the standard or the study treatment. Patient preference was compared between the standard and the study treatment with a Chi-Square test for equal proportion

4. Other Pre Specified Outcome: Incidence of Ocular Adverse Events Reported Throughout the Study
Description: A targeted physical examination was performed at all visits and monitoring for ocular and systemic adverse events occurred throughout the study
Time Frame: From Visit 2 (baseline) to Visit 3 (week 4)
Population: Patiens with symmetrical bilateral posterior blepharitis who applied treatment at least once in one eye.
  One patient reported a treatment-emergent systemic adverse event, i.e. "Suspected colon cancer" of mild severity that led to permanent treatment discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment | Standard Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Eyes with Serious Ocular Adverse Event | 0 | 0
  Eyes with Ocular Adverse Event | 8 | 7
Statistical Analysis 1: Comparison: Study Treatment vs Standard Treatment; Test type: Other; p = 0.7353, Chi-squared; The incidence of all the treatment-emergent systemic Adverse Events recorded in the eCRF was presented overall at patient level; the incidence of all the treatment-emergent ocular Adverse Events recorded in eCRF was presented by treatment group at eye level. Incidence of treatment-emergent ocular Adverse Events was compared between treatment groups by means of a Chi-square test

5. Other Pre Specified Outcome: Compliance to Treatment Evaluated by Counting the Applications (Wet Wipes) to Each Eyes
Description: Adherence to treatment was evaluated at Visit 3 by counting given wipes/gauze and unused/lost/damaged wipes/gauze.
  The compliance to treatment was evaluated by counting given wipes/gauze and unused/lost/damaged wipes/gauze. The following formula was applied:
  (Given wipes/gauze - (sum of unused/lost/damaged wipes/gauze)) / Expected number of wipes/gauze used) x 100. Where the "given wipes/gauze" were 60 and the "expected number of wipes/gauze used" were 2 per days per 4 weeks = 56.
Time Frame: From Visit 2 (baseline) to Visit 3 (week 4)
Population: Patiens with symmetrical bilateral posterior blepharitis who applied treatment at least once in one eye.
Measure: Mean (Standard Deviation); unit: percentage of Application (Wet Wipes)
Arm/Group | Study Treatment | Standard Treatment
Number analyzed (Participants) | 18 | 18
percentage of Application (Wet Wipes) | 96.1 (8.8) | 94.2 (9.5)

ADVERSE EVENTS:
Time Frame: from baseline to week 4
Description: The patient will be given a diary on which to record the application of all morning and evening treatments, as well as any adverse events occurred. The diary is to be returned at Visit 3 for review
Arm/Group | Study Treatment | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/18 | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=18) | Standard Treatment (N=18)
Dry eye (Eye disorders) | 3 | 3
Ocular pain (Eye disorders) | 4 | 2
Irritation (Eye disorders) | 2 | 2
Itching or discomfort (Eye disorders) | 3 | 2
Increased lacrimation (Eye disorders) | 2 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 1
Ocular secretions (Eye disorders) | 1 | 1
Crusts on eyelid margins (Eye disorders) | 1 | 1
Blurred vision (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 2 | 1
Purulent discharge (Eye disorders) | 1 | 0
Madarosis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03301844/Prot_SAP_000.pdf